CLINICAL TRIAL: NCT06478615
Title: Coring Out Fistulectomy With Closure of Internal Sphincter Opening Versus Lay Open Fistulotomy and Primary Sphincter Repair in Transsphincteric Perianal Fistula; A Prospective Randomized Comparative Study
Brief Title: Coring Out Fistulectomy With Closure of Internal Sphincter Opening Versus Lay Open Fistulotomy and Primary Sphincter Repair in Transsphincteric Perianal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ali Ahmed, Assistant Lecturer of General Surgery, Faculty of Medicine, Ain Shams University, Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30/10/2022
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Coring Out; Fistulectomy; Internal Sphincter; Lay Open Fistulotomy; Sphincter Repair; Transsphincteric Perianal Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coring out Fistulectomy with Closure of Internal Sphincter Opening (Experimental): Patients underwent coring out fistulectomy with closure of internal sphincter opening
  Interventions: Procedure: Coring out Fistulectomy with Closure of Internal Sphincter Opening
- Lay Open Fistulotomy and Primary Sphincter Repair (Experimental): Patients underwent lay open fistulotomy and primary sphincter repair
  Interventions: Procedure: Lay Open Fistulotomy and Primary Sphincter Repair

INTERVENTIONS:
Procedure: Coring out Fistulectomy with Closure of Internal Sphincter Opening — The patient was laid in the lithotomy position. Skin preparation and draping were done. Normal saline irrigation was performed. The anal canal was sufficiently dilated to permit the introduction of a self-retaining retractor. With H2O2 injection into the fistula tract, the internal opening and tract of the fistula will be identified. The incision was made around the external opening, and the tract was all cored out along the tract from the external opening to the internal sphincter. Meticulous hemostasis will be performed, stay suture by PDS 4/0 around fistiolous opening at the internal sphincter, excision of fistulous tract above stay suture, then closure of internal sphincter defect by PDS 3/0. Anal packing with 4 × 4 epinephrine gauze and sterile protective dressing was performed. After the operation, a stool softener and pain controller were prescribed, and patients were discharged.
  Arms: Coring out Fistulectomy with Closure of Internal Sphincter Opening
Procedure: Lay Open Fistulotomy and Primary Sphincter Repair — Patients were put in a lithotomy position and the skin was then draped. After identification of the external fistula orifice probing of the fistula tract with identification of the fistulous tract and internal orifice with H2O2 injection into the fistula tract. The fistula was laid open and fistulectomy was then conducted and dissected with diathermy cautery help. Then Primary repair of the sphincter with PDS 3/0 with proper hemostasis using coagulation diathermy.
  Arms: Lay Open Fistulotomy and Primary Sphincter Repair

SUMMARY:
This study aimed to compare the surgical outcomes of coring out fistulectomy with the closure of internal sphincter opening versus lay open fistulotomy (modified LIFT) and lay open fistulotomy and primary sphincter repair in trans-sphincteric perianal fistula

DETAILED DESCRIPTION:
Fistula-in-ano is a common medical problem affecting thousands of patients annually. Symptoms generally affect quality of life significantly, and they range from minor discomfort and drainage with resultant hygienic problems to sepsis. Different classifications have been put forward which categorize these Fistula into low or high simple or complex, or according to their anatomy inter-sphincteric, trans-sphincteric, and supra- sphincteric or extra-sphincteric.

Conventional laying-open technique in high perianal fistula may involve sacrifice of part or whole of the sphincter muscle impairing continence. A transposition technique for the management of high anal and anorectal fistulae is described by Mann and Clifton in 1985. The method involves re-routing the extrasphincteric portion of the track into an intersphincteric position with immediate repair of the external sphincter.

Coring-out fistulectomy is a type of sphincter-preserving procedure that enables accurate resection of the fistula tract alone and thus reduces the possibility of missing a secondary tract

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I, II.
* Fistula in ano, Trans-sphincteric type

Exclusion Criteria:

* Patients with low perianal fistula.
* Recurrent perianal fistula.
* Associated anal conditions such as (piles, anal fissures, and rectal prolapse).
* Patients with inflammatory bowel disease or tuberculosis.
* Patients with acute perianal abscess.
* Patients with major incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrence of perianal fistula | 3 months postoperatively
  Incidence of recurrence of perianal fistula was recorded and confirmed when an anal fistula or abscess is observed on any previously healed wound for 3 months.

SECONDARY OUTCOMES:
Incidence of stool incontinence | 3 months postoperatively
  Incidence of stool incontinence was recorded for 3 months.
Healing time | 3 months postoperatively
  Healing was defined as cicatrization of all wounds without discharge at 3 months
Length of hospital stay | 1 week postoperatively
  Length of hospital stay was recorded from admission till discharge from hospital.
Complications | 3 months postoperatively
  Complications such as (blood loss, pain, bleeding, discharge, urinary retention, urgency, wound infection) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.